CLINICAL TRIAL: NCT03390777
Title: Plasma Rich in Growth Factors for Treatment of Medication Related Osteonecrosis of the Jaw: a Multicenter, Randomized, Clinical Trial
Brief Title: Plasma Rich in Growth Factors for Treatment of Medication Related Osteonecrosis of the Jaw
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Collaborators: NYU College of Dentistry (Other); Universidade da Coruña (Other)
Responsible Party: Principal Investigator, Oreste Iocca, DDS, MD, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 26122017
Record Dates: First submitted 2017-12-26; First posted 2018-01-04 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Osteonecrosis Due to Drugs, Jaw
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- surgery only (Active Comparator): Surgery consisting in debridement/removal of affected tissue/s will be performed.
  Interventions: Procedure: surgery
- surgery and PRGF (Active Comparator): Surgery consisting in debridement/removal of affected tissue/s will be performed. Platelet Rich Growth Factor (device) will be produced by a venous blood sampling of the patient and applied to the treated area
  Interventions: Device: PRGF after surgery

INTERVENTIONS:
Procedure: surgery — surgery without the use of prgf
  Arms: surgery only
Device: PRGF after surgery — surgery and application of PRGF
  Arms: surgery and PRGF

SUMMARY:
Medication related Osteonecrosis of the Jaw (MRONJ) consists of progressive destruction of bone in the maxillofacial area. It is an established complication which occurs in patients who take two main classes of antiresorptive drugs: Bisphosphonates (BP) and Denosumab.

PRGF is a autologous platelet-enriched plasma obtained from the patient's own blood. It contains proteins that can influence and promote cell recruitment and its beneficial effect could consist in improving bone and soft tissue healing. These benefits are likely to apply to MRONJ surgery, as it is suggested by small retrospective or prospective case series.

This is a randomized, multi center study comparing the outcomes of surgery alone and PRGF plus surgery in patients requiring surgical treatment for MRONJ.

To assess the superiority of surgery plus PRGF compared to surgery alone in patients treated for MRONJ. Primary endpoint for this scope is a composite of clinical or radiological recurrence rate of disease during a 12 months post-operative period.

Secondary endpoints are: a) morbidity, defined as nerve injury, bleeding, vascular or wound complications. b) post- and peri-operative pain defined by the treated subjects according to a standardized VAS score c) quality of life (QoL) defined by a standardized scale.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be candidates for surgical treatment for MRONJ at stage 2 or 3.
* Subjects must be >18 and <80 years of age
* Subjects must sign a informed consent prior to randomization and must agree to return to scheduled follow-up visits

Exclusion Criteria:

* Subject has inability to understand and cooperate with the study procedures or provide informed consent
* Subject has bleeding diathesis or coaugolapthy, or will refuse autologous blood sampling
* Subject had a cardiovascular event in the past 30 days
* Subject has any condition that limits their anticipated survival to less than 3 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
recurrence of disease | 12 months
  clinical or radiological recurrence rate of disease during a 12 months post-operative period

SECONDARY OUTCOMES:
morbidity | 12 months
  nerve injury, bleeding, vascular or wound complications
post- and peri-operative pain | 1 week
  defined by the treated subjects according to a standardized Visual Analog Scale (VAS) score which will be used to define the pain in this way: the patient will assign a value to the experienced pain that goes from 0 no pain to 10 the worst pain the patient can imagine.
quality of life (QoL) | 12 months
  defined by a standardized scale developed by the who and whose details can be on the who website http://www.who.int/mental_health/publications/whoqol/en/

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared and evaluated upon requests
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Derived] Beth-Tasdogan NH, Mayer B, Hussein H, Zolk O, Peter JU. Interventions for managing medication-related osteonecrosis of the jaw. Cochrane Database Syst Rev. 2022 Jul 12;7(7):CD012432. doi: 10.1002/14651858.CD012432.pub3. PMID 35866376